CLINICAL TRIAL: NCT05864105
Title: A Phase II Study to Evaluate the Efficacy, Safety and Pharmacokinetics of PM8002 Injection in Combination With Standard Chemotherapy as First Line Therapy in Unresectable Hepatocellular Carcinoma
Brief Title: PM8002 in Combination With Chemotherapy as First Line Therapy in Hepatocellular Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biotheus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM8002 -B006C-HCC-R
Record Dates: First submitted 2023-05-09; First posted 2023-05-18 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: PD-L1/VEGF; FOLFOX-4
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Folfox protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PM8002+FOLFOX-4 (Experimental): PM8002 20mg/kg Q2W day 1: oxaliplatin [85 mg/m2, 2-h infusion] plus leucovorin [200 mg/m2, 2-h infusion], followed by 5-fluorouracil [400 mg/m2, intravenous bolus; 600 mg/m2, 22-h infusion]; day 2: leucovorin [200 mg/m2, 2-h infusion], followed by 5-fluorouracil [400 mg/m2, intravenous bolus; 600 mg/m2, 22-h infusion]
  Interventions: Biological: PM8002; Drug: FOLFOX regimen

INTERVENTIONS:
Biological: PM8002 — PM8002 20mg/kg Q2W
Drug: FOLFOX regimen — day 1: oxaliplatin [85 mg/m2, 2-h infusion] plus leucovorin [200 mg/m2, 2-h infusion], followed by 5-fluorouracil [400 mg/m2, intravenous bolus; 600 mg/m2, 22-h infusion]; day 2: leucovorin [200 mg/m2, 2-h infusion], followed by 5-fluorouracil [400 mg/m2, intravenous bolus; 600 mg/m2, 22-h infusion]

SUMMARY:
This is a multicenter, single-arm, open-label phase II study to evaluate the efficacy and safety of PM8002 in combination with chemotherapy in the first-line treatment of subjects with inoperable HCC.

DETAILED DESCRIPTION:
PM8002 is a Bispecific Antibody Targeting PD-L1 and VEGF.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in clinical study; fully understand the study and sign informed consent voluntarily; willing to follow and able to complete all test procedures;
2. Male or female aged >= 18 years;
3. HCC diagnosed by pathology or clinical;
4. BCLC stage C or B (unresectable or/and not suitable for local therapy);
5. Child-Pugh score <= 7;
6. ECOG performance status of 0 or 1.

Exclusion Criteria:

1. Histological diagnosis of fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC;
2. Symptomatic CNS metastases, not suitable for the study assessed by investigator;
3. Evidence of major coagulopathy or other obvious risk of bleeding;
4. Unable to accept enhanced imaging examination (CT or MRI) for any reason;
5. History of severe allergic disease, severe allergy to drugs or known allergy to any component of the drug in this study;
6. Human immunodeficiency virus infection or known acquired immunodeficiency syndrome;
7. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
8. Known history of alcohol abuse, psychotropic drug abuse or drug abuse;
9. Patients with psychiatric disorders or poor compliance;
10. Women who are pregnant or breastfeeding;
11. The condition of the subject, as determined by the investigator, may increase the risk of after study treatment, or may cause confusion about the interpretation of the toxic reaction and AE;
12. Other conditions lead to inappropriate to participate in this study as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Up to approximately 2 years
  Objective response rate (ORR) is the proportion of subjects with complete response (CR) or partial response (PR), based on RECIST v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Jieer Ying, Principal Investigator — Cancer Hospital of The University of Chinese Academy of Sciences
Locations (9):
- China (9):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Hospital of Jilin University, Changchun, Jilin
  - Cancer Hospital of The University of Chinese Academy of Sciences, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Jinhua Municipal Centeral Hospital Medical Group, Jinhua, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
The data will be published or presented for publications (poster, abstract, articles or papers) or any presentations.